CLINICAL TRIAL: NCT06045299
Title: A Multi-Center, Randomized, Double-Masked, Placebo-Controlled Phase 3 Evaluation of the Efficacy and Safety of LNZ101 and LNZ100 for the Treatment of Presbyopia
Brief Title: Evaluation of the Efficacy and Safety of LNZ101 and LNZ100 for the Presbyopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: LENZ Therapeutics, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JX07001; CTR20232913 (Other: China CDE clinical trial registration)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-09

CONDITIONS: Presbyopia; Near Vision; Miosis; Eye Diseases
Keywords: Presbyopia; Pharmaceutical Solutions; Opthalmic Solutions; Eye Drops; Miotic
MeSH Terms: conditions — Presbyopia; Myopia; Miosis; Eye Diseases | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LNZ101 (Aceclidine/Brimonidine) ophthalmic solution (Experimental): Enrolled subjects will be randomized to receive LNZ101, LNZ100, or placebo bilaterally once a day. Subjects will be instructed to dose 2 drops in both eyes (OU) (1 drop followed by 2 minutes later, another drop). Subjects will dose for 168 days.
  Interventions: Drug: Aceclidine+Brimonidine combination ophthalmic solution
- LNZ100 (Aceclidine) ophthalmic solution (Experimental): Enrolled subjects will be randomized to receive LNZ101, LNZ100, or placebo bilaterally once a day. Subjects will be instructed to dose 2 drops in both eyes (OU) (1 drop followed by 2 minutes later, another drop). Subjects will dose for 168 days.
  Interventions: Drug: Aceclidine ophthalmic solution
- Placebo (Vehicle) ophthalmic solution (Placebo Comparator): Enrolled subjects will be randomized to receive LNZ101, LNZ100, or placebo bilaterally once a day. Subjects will be instructed to dose 2 drops in both eyes (OU) (1 drop followed by 2 minutes later, another drop). Subjects will dose for 168 days.
  Interventions: Drug: Placebo (Vehicle) ophthalmic solution

INTERVENTIONS:
Drug: Aceclidine+Brimonidine combination ophthalmic solution — Aceclidine+Brimonidine combination ophthalmic solution
  Other Names: LNZ101
  Arms: LNZ101 (Aceclidine/Brimonidine) ophthalmic solution
Drug: Aceclidine ophthalmic solution — Aceclidine ophthalmic solution
  Other Names: LNZ100
  Arms: LNZ100 (Aceclidine) ophthalmic solution
Drug: Placebo (Vehicle) ophthalmic solution — Placebo (Vehicle) ophthalmic solution
  Arms: Placebo (Vehicle) ophthalmic solution

SUMMARY:
A Multi-Center, Randomized, Double-Masked, Placebo-Controlled Phase 3 Evaluation of the Efficacy and Safety of LNZ101 and LNZ100 for the Treatment of Presbyopia

DETAILED DESCRIPTION:
A multicenter, randomized, double-masked, placebo-controlled efficacy and safety study . To evaluate the efficacy and safety of LNZ101 (Aceclidine 1.75%/Brimonidine 0.08%)/LNZ100 (Aceclidine 1.75%) compared with placebo for the treatment of presbyopia.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent prior to any study procedure being performed;
2. Be able and willing to follow all instructions and attend all study visits;
3. Be 45-75 years of age of either sex at Visit 1;
4. Have +1.00 to -4.00 diopter (D) of sphere calculated in minus cylinder in both eyes determined by manifest refraction documented at Visit 1;
5. Have ≤2.00 D of cylinder (minus cylinder) in both eyes determined by manifest refraction documented at Visit 1;
6. Have +1.00 D to -4.00 D manifest refraction spherical equivalent（MRSE）of Spherical equivalent (SE) determined by manifest refraction documented at Visit 1.
7. Be presbyopic as determined at Visit 2 baseline

Exclusion Criteria:

1. Be a female of childbearing potential who is currently pregnant, nursing, or planning a pregnancy;
2. Have known contraindications or sensitivity to the use of any of the study medications or their components;
3. Have an active ocular infection at Visit 1 or at Visit 2 (bacterial, viral, or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation (e.g., moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis, scleritis, uveitis) in either eye;
4. Have moderate or severe dry eye at Visit 1, assessed by corneal fluorescein staining;
5. Have clinically significant abnormal lens findings (e.g., cataract) including early lens changes and/or any evidence of a media opacity during dilated slitlamp biomicroscopy and fundus exam documented within 3 months of Visit 1 or at Visit 1;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Best-corrected distance visual acuity (BCDVA) at 40 cm | 3 hours post-treatment in the study eye at Visit 2 (Day 1）
  Percentage of subjects who achieve a 3-line (15-letter) or greater improvement from baseline in the measurement of monocular BCDV at 40 cm and no loss in BCDVA ≥ 5 letters (ETDRS chart at 4 m)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Sun, Study Director — Corxel Pharmaceuticals
Locations (19):
- China (19):
  - Eye Hospital, Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Ineye Hospital of Chengdu University of TCM, Chengdu
  - Dalian N0.3 people's hospital, Dalian
  - Guang Zhou Aier eye Hospital, Guangzhou
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Affiliated Eye Hospital, Shandong University of Traditional Chinese Medicine, Jinan
  - Shanghai Eye Disease Prevention and Treatment Center, Shanghai
  - Tongji Hospital Of Tongji University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School Of Medicine, Shanghai
  - Shanxi Eye Hospital, Taiyuan
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital, Tianjin
  - Wuhan Aier Eye Hospital, Wuhan
  - Xi'An People's Hospital, Xi'an
  - Henan Eye Hospital & Henan Institute, Zhengzhou